CLINICAL TRIAL: NCT01690325
Title: Molecular Imaging for Response Assessment of Bevacizumab + Docetaxel as Neoadjuvant Chemotherapy in Primary Breast Cancer
Brief Title: Imaging for Response Assessment of Neoadjuvant Chemotherapy in Primary Breast Cancer (GALADON)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Therapy of HER2+ patients according to protocol was no longer appropriate. Patient enrolment behind planned schedule and challenges of site performance
Sponsor: West German Study Group (Other)
Collaborators: Roche Pharma AG (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSG-AM05
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant chemotherapy; Neoadjuvant cytotoxic-antiangiogenic therapy; Bevacizumab; PET
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Trastuzumab; Bevacizumab; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel, Avastin, Herceptin; adjuv. Epirubicin, Cyclophos. (Experimental): Arm A: Neoadjuvant: 6 cycles of Docetaxel every 21 days together with 6 cycles of Avastin and Herceptin; Adjuvant: 4 cycles of Epirubicin and Cyclophosphamid every 21 days together with 12 cycles of Herceptin every 21 days.
  Interventions: Drug: Docetaxel; Drug: Trastuzumab; Drug: Bevacizumab; Drug: Epirubicin; Drug: Cyclophosphamid
- Docetaxel, Avastin; adjuvant Epirubicin, Cyclophosphamid (Experimental): Arm B: neoadjuvant: 6 cycles of Docetaxel and Avastin every 21 days. Adjuvant: 4 cycles of Epirubicin and Cyclophosphamid every 21 days.
  Interventions: Drug: Docetaxel; Drug: Bevacizumab; Drug: Epirubicin; Drug: Cyclophosphamid

INTERVENTIONS:
Drug: Docetaxel
Drug: Trastuzumab
  Other Names: Herceptin
  Arms: Docetaxel, Avastin, Herceptin; adjuv. Epirubicin, Cyclophos.
Drug: Bevacizumab
  Other Names: Avastin
Drug: Epirubicin
Drug: Cyclophosphamid

SUMMARY:
The GALADON trial is a diagnostic and interventional study in which different molecular imaging methods as Positon Emission Tomography (PET), different kind of Magnetic Resonance Imaging - methods (MRI, DWI and DCE-MRI) will be compared with common imaging methods (mammography, ultrasound) to see if there can detect an early response to a combined neoadjuvant therapy with bevacizumab and docetaxel in patients with locally advanced breast cancer. Neoadjuvant chemotherapy (this means patients were treated before the tumor was removed by surgery) with a drug like trastuzumab (monoclonal antibody) which is target to the Her2-protein is much more powerful than with chemotherapy alone because it is normalizing the blood supply and improves tumor delivery of conventional chemotherapy like docetaxel. The HER2 protein is only available in about 30 % of breast cancer types. bevacizumab is another humanized monoclonal antibody like trastuzumab but is effective not only in patients with an positive HER2 status and in combination with trastuzumab it may emphasize the effect in reduction of tumor growth. Bevacizumab is approved in advanced disease, but no major neoadjuvant data available so far for primary breast cancer. As the therapy with monoclonal antibody regimes are expensive and may cause severe side effects predictive factors to select patients who will benefit from such highly specific drugs before therapy start would be medically and economically highly valuable. In this study the efficacy of combined neoadjuvant chemotherapy with bevacizumab, trastuzumab and docetaxel in Arm A and bevacizumab and docetaxel in Arm B should be evaluated and the predictive impact of different imaging methods for tumor response should be shown.

ELIGIBILITY:
Inclusion Criteria:

Arm A / Arm B

* Age ≥ 18 years and ≤ 65 years
* Female
* Operable, locally advanced primary breast cancer (≥ cT2, N0 or N+, M0) histologically confirmed by core biopsy
* Histologically confirmed unilateral, solitaire breast cancer
* Patients who are candidates for neoadjuvant chemotherapy according to AGO guidelines (www.ago-online.de) with unifocal lesion
* HER2 positive disease (IHC 3+ and/or FISH positive)or
* HER2 negative disease (IHC 0/1+, IHC 2+ and/or FISH negative)
* Baseline LVEF ≥ 55% (measured by MUGA or echocardiography) according to institution specific norm
* Informed consent for clinical trial including analysis of predictive imaging tests and biomarkers
* Clinically or by imaging (mammogram, MRI or US) assessed breast cancer ≥ 2 cm or inflammatory breast cancer with bi-dimensional measurable lesion independent of nodal status
* Negative pregnancy test (urine or serum) within 7 days prior to registration if patient is premenopausal with intact reproductive organs and if patient is less than one year after menopause
* ECOG Performance status 0-2
* Adequate organ function for cytotoxic chemotherapy
* Adequate renal function including Serum creatinine ≤ ULN, Measured or calculated creatinine clearance > 60 ml/min
* Urine dipstick for proteinuria < 2+. In case of ≥ 2+ proteinuria on dipstick urinalysis, a 24-hour urine collection must be performed and protein per 24 hours must be ≤ 1.0 g
* Absolute neutrophil count ≥ 1500 cells/μl, platelet count ≥ 100,000 cells/μl
* Bilirubin ≤ ULN; ALT or AST ≤ 1.5 x ULN, and alkaline phosphatase < 2.5 x ULN
* Patients must be available and compliant for treatment and follow-up

Exclusion Criteria:

Arm A / Arm B

* Evidence of distant metastases by clinical or imaging diagnosis
* Multifocal primary tumour, defined as histologically confirmed tumour-manifestations within different quadrants; distance ≥ 4 cm
* Pre-existing motor or sensory neuropathy of a severity ≥ grade 2 NCI criteria
* Previous breast cancer
* Prior malignancy with a disease-free survival of < 5 years
* Prior malignancy which has not been curatively treated
* Inflammatory breast cancer without bi-dimensional measurable lesion
* Prior systemic therapy for cancer
* Previous therapy with trastuzumab or other anti-HER2 agent (for HER2+ tumors)
* Previous therapy with bevacizumab or other anti-VEGF agent
* Patients with immunosuppressive therapy
* Pregnant or lactating women
* Women of childbearing potential not using highly effective birth control.
* Patients with known hypersensitivity reactions to the compounds or incorporated substances of trastuzumab or its constituents (for HER2+ tumors).
* Patients with known hypersensitivity reactions to the compounds or incorporated substances of bevacizumab or its constituents.
* Invasive malignancy which could affect compliance with the protocol or interpretation of results.
* Other serious illness or medical condition including:

  * Known or suspected congestive heart failure (>NYHA I) and/or coronary heart disease
  * Angina pectoris requiring antianginal medication
  * Previous history of myocardial infarction
  * Evidence of transmural infarction on ECG
  * Un- or poorly controlled arterial hypertension (i.e. BP >150/100 mmHg under treatment with two antihypertensive drugs)
  * Rhythm abnormalities requiring permanent treatment
  * Clinically significant valvular heart disease
  * Patients with dyspnoea at rest due to malignant or other disease or who require supportive oxygen therapy
  * Active serious uncontrolled infections
  * Poorly controlled diabetes
  * History of hypertensive crisis or hypertensive encephalopathy
  * History of TIA or CVA
  * History of any arterial thrombotic event within 12 months before randomization
* Inadequate bone marrow, hepatic and renal functions as evidenced by the following:
* Neutrophil count of < 1500, platelet count of < 100,000/µL
* Haemoglobin < 10 g/dL
* Serum total bilirubin > ULN (except for patients with clearly documented Gilbert's syndrome)
* ALT or AST > 1.5 x ULN
* Alkaline phosphatase > 2.5 x ULN, serum creatinine > ULN
* Concurrent treatment with any other anti-cancer therapy
* No informed consent for analysis of predictive imaging tests and biomarkers
* Contraindications against MRI: Cardiac pacemakers, other forms of medical or biostimulation implants, ferromagnetic foreign bodies or metallic implants (e.g. surgical protheses, aneurysm clips), implanted insulin pumps, valvular implants, allergy to contrast agent, renal insufficiency, claustrophobia
* Active peptic ulcer, incomplete wound healing or unhealed bone fracture
* Previous thromboembolic events, known hemorrhagic diathesis, coagulopathy with increased bleeding risk, or treatment with anticoagulants. Current or recent (within 10 days of first dose of bevacizumab) use of acetalic acid (> 325 mg/day) or clopidogrel (> 75 mg/day)
* Disease significantly affecting gastrointestinal function, e.g. malabsorption syndrome, resection of the stomach or small bowel, ulcerative colitis; abdominal fistula, intra-abdominal abscess within 6 months of enrolment or gastrointestinal perforation
* Major surgery within the last 28 days or anticipation of the need for major surgery during study treatment with bevacizumab. No minor surgeries including insertion of an indwelling catheter within 24h prior to registration.
* Concurrent treatment with other experimental drugs; participation in another clinical trial with any investigational drug within 30 days prior to study entry
* Chronic daily treatment with corticosteroids (dose of > 10 mg/day methylprednisolone equivalent) (excluding inhaled steroids).
* Patients with a history of hypersensitivity reaction to docetaxel or to drugs formulated with polysorbate 80

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Rate of pathological complete response (pCR) following neoadjuvant therapy in group A and group B | about 18 weeks (start of neoadjuvant chemotherapy until surgery)
  To determine efficacy of cytotoxic-antiangiogenic neoadjuvant therapy in primary breast cancer: bevacizumab+trastuzumab+docetaxel fro group A (HER2 positive) or bevacizumab+docetaxel for group B (HER2 negative) using pathological complete response (pCR) as the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Harbeck, Prof. Dr. med., Principal Investigator — Head of Breast Centre, University of Munich, Grosshadern Hospital, Germany
Locations (1):
- Breast Centre, University of Munich, LMU, Munich, Bavaria, Germany